CLINICAL TRIAL: NCT02210988
Title: Evaluating the Therapeutic Effect of Acupuncture on Acute Ischemic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cathay General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGHIRBCT-P-100002
Record Dates: First submitted 2014-07-14; First posted 2014-08-07 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2014-08

CONDITIONS: Acute Stroke
Keywords: Acupuncture therap; Acute stroke; Randomized controlled trials
MeSH Terms: conditions — Stroke | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- acupuncture (Experimental): The acupuncture treatment for the intervention group was provided once daily for 2 weeks.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — Intervention with acupuncture

SUMMARY:
The investigators design a randomized, single blinded, control study to evaluate the therapeutic effect of acupuncture in acute ischemic stroke patients:

DETAILED DESCRIPTION:
Acupuncture therapy in traditional Chinese medicine has been verified in many disease by thousands years. Due to the feasible and relatively safe in acupuncture management, now the west countries had been well document about acupuncture in medicine. The acupuncture therapy applied in post stroke functional recovery has been considered as more benefit than physical therapy only to post stroke rehabilitation. However, the effect of combined acupuncture therapy with standard management in acute stroke patient still remains unknown. The aim of this study is to evaluate the therapeutic effect of acupuncture in acute ischemic stroke patients. The prospective study was designed as a randomized, single blinded, control trial. We collected newly onset of acute ischemic stroke patient without underling systemic major illness, and randomized assign the collected patients into two groups as experimental (acupuncture)group and normal control group. The two groups both treat with routine western medicine as standard stroke therapy. The outcome measurement will evaluate by the changes from baseline at one and three months. The assessed scales including NIH stroke scale, the Barthel index, the Functional Independence Measure score, the Fugl-Meyer Assessment, and the Modified Rankin Scale. We compared the all variable measurements to see if any benefit from acupuncture group than the control group.

ELIGIBILITY:
Inclusion Criteria:

* newly onset of acute ischemic stroke,Exclusion Criteria:
* without underling systemic major illness

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
National Institute of Health Stroke Scale | the fourth week
Fugal-Mayer Assessment | The fourth week
Functional Independent Measure | The fourth week

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale | The three months after admission
Barthel index | The three month after admission
Modified Rankin Scale | The three after admission

OTHER OUTCOMES:
Number of Participants with Adverse Events | The two week
  Adverse events was monitored in each acupuncture maneuver and post therapeutic course two weeks later.

REFERENCES:
- [Derived] Liu CH, Hsieh YT, Tseng HP, Lin HC, Lin CL, Wu TY, Lin SH, Tsao SH, Zhang H. Acupuncture for a first episode of acute ischaemic stroke: an observer-blinded randomised controlled pilot study. Acupunct Med. 2016 Oct;34(5):349-355. doi: 10.1136/acupmed-2015-010825. Epub 2016 Apr 19. PMID 27095698